CLINICAL TRIAL: NCT01513811
Title: High Dose of Itopride: a Valid Adjuvant for Bowel Preparation in Patients With Chronic Constipation
Brief Title: Itopride as an Adjuvant for Bowel Preparation in Patients With Chronic Constipation is Effective
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Xiaobo Li, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rjyyxhk0906
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Constipation
Keywords: bowel preparation; constipation; polyethylene glycol; itopride
MeSH Terms: conditions — Constipation | interventions — itopride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- group PEG (Active Comparator): This group is set as a control group and received 2 packets of Polyethylene glycol electrolyte solutions on the morning of the examination day as us we usually done.
  Interventions: Drug: Polyethylene glycol electrolyte solutions
- group PEG+Itp (Active Comparator): Patients in group were assigned to itopride half hour before administration of lavage solution in the morning of examination day.
  Interventions: Drug: Itopride and Polyethylene glycol electrolyte solutions
- group PEG+4Itp (Active Comparator): Patients in this group received itopride three times 24 hours before the examination day and another time 30 min before administration of lavage solution.
  Interventions: Drug: itopride and polyethylene glycol electrolyte solutions

INTERVENTIONS:
Drug: Polyethylene glycol electrolyte solutions — Patients received 2 packets of polyethylene glycol electrolyte solutions(PEG-E) without itopride.PEG-E was dissolved in 2 L of water. Patients were instructed to drink PEG solution 200ml every 10 min consumed the total 2 L solution in 2 hours.6 hours later, the colonoscopy was performed.
  Other Names: PEG-E
  Arms: group PEG
Drug: Itopride and Polyethylene glycol electrolyte solutions — Patients were assigned to itopride 150mg, then 30 min later they were given 2 packets of polyethylene glycol electrolyte solutions(PEG-E). PEG-E was dissolved in 2 L of water. Patients were instructed to drink PEG solution 200ml every 10 min consumed the total 2 L solution in 2 hours. 6 hours later, the colonoscopy was performed.
  Other Names: PEG-E; Itopride hydrochloride
  Arms: group PEG+Itp
Drug: itopride and polyethylene glycol electrolyte solutions — Patients received itopride 150mg t.i.d(7am、12am、8pm) 24 hours before the examination day and another 150mg 30min before administration of polyethylene glycol electrolyte solutions(PEG-E).Two packets of PEG-E were dissolved in 2 L of water. Patients were instructed to drink PEG solution 200ml every 10 min and consumed the total 2 L solution in 2 hours. 6 hours later, the colonoscopies were performed.
  Other Names: PEG-E; itopride hydrochloride
  Arms: group PEG+4Itp

SUMMARY:
Bowel preparation is a major determinant of colonoscopy and colorectal surgery. Polyethylene glycol electrolyte solutions (PEG-E) are the most commonly used laxatives in China. However, a significant number of patients, especially those constipated patients, failed colonoscopies due to poor bowel cleaning. Inadequate preparation may also lead to missed colonic lesions. The study is based on the hypothesis: itopride hydrochloride, a prokinetic agent, its dual role as dopamine D2 receptor antagonism and acetylcho-linesterase inhibition make it an appropriate adjuvant for bowel preparation. It was reported to promote colonic peristalsis, shorten colonic transit time and accelerate propulsion of colonic luminal contents through inhibition of M3 receptor and dopamine D2 receptors in vitro and in vivo. So this study is to determine the efficacy, tolerance and safety of high dose of itopride, when given in different times before administration of PEG-E, for colonic preparation in patients with chronic constipation.

DETAILED DESCRIPTION:
Colonoscopy is a reliable procedure for the investigation of colonic and distal terminal ileum disease. The diagnostic accuracy of colonoscopy is dependent on visualization of the colonic mucosa; hence an appropriate bowel preparation is essential for the examination. Despite multiple lavage were used throughout the years, the suboptimal cleaning level have been reported vary from 10% to more than 20% and up to one-third of incomplete or failed colonoscopies can be ascribed to poor bowel preparation. So it is important for us to search a new regimen for bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected colonic disease and suffered from chronic constipation were referred for colonoscopy and enrolled in the study. Chronic constipation was diagnosed on the basis of Rome III criteria.Suspected colonic disease was deﬁned as:

  * recent change of bowel habits;
  * obscure GI bleeding (hemafecia, melena or positive fecal occult blood test);
  * obscure abdominal pain;
  * weight loss;
  * positive ﬁndings in the colon on GI imaging;
  * serological test referred to colorectal cancer such as CEA elevated obviously;
  * family history of colorectal cancer or adenomatous polyps.

Exclusion Criteria:

* usage of prokinetic agents such as itopride, mosapride within 4 weeks and tricyclic antidepressants 8 weeks prior to entering the protocol;
* known allergies or other contraindication to PEG or itopride;
* a history of abdominal surgery or bowel obstruction;
* pregnant or lactating;
* conditions associated with severe cardiac, hepatic, or renal impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
the quality of bowel preparation | the day of colonoscopy examination
  the Boston Bowel Preparation Scale (BBPS): the colon was divided into 3 broad segments: the right side (the cecum and ascending colon), the middle section (the hepatic ﬂexures, transverse colon and splenic ﬂexures), and the left side of the colon (the descending colon, sigmoid colon, and rectum). Each region of the colon receives a score from 0 to 3 as summarized in table 1, score 0 was considered poor preparation while score 3 indicated good cleaning quality. And these segment scores are summed for a total BBPS score ranged from 0 to 9.

SECONDARY OUTCOMES:
intestinal bubble scale | the day of colonoscopy examination
  The scores of intestinal bubble were categorized into three levels: 0, no or nearly no bubble present; 1, small amounts of bubbles that could be washed away easily; 2, multiple collections of bubbles that could be washed away with volumes of water.
time of examination | the day of examination
  Time of examination includes caecal intubation time and withdrawal time. Caecal intubation time deﬁned as the time passing the colonoscope to the ileocaecal valve. Withdrawal time deﬁned as the time withdrawing from ileocaecal junction to anus.
times of defecation | the day before and the day of examination
  The times of defecation during the preparation were obtained and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Li X B, M.D., Ph.D., Study Chair — Shanghai Jiao-Tong University School of Medicine Renji Hospital
Locations (1):
- Shanghai Jiao-Tong University School of Medicine Renji Hospital, Shanghai, Shanghai Municipality, China